CLINICAL TRIAL: NCT04161625
Title: Evaluation of Reach, Effects and Cost Effectiveness of a Fall Preventive Intervention Including a mHealth Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SafeStepReach
Record Dates: First submitted 2019-10-09; First posted 2019-11-13 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Accidental Falls
Keywords: Prevention and control; Exercise therapy/methods*; Aged 70 and over; Smartphone; Computers handheld; Motivation; Behaviour change; Postural balance; Health behaviour; mHealth; eHealth; Digital health; Self-management; Re-aim
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: This is a pragmatic clinical trial evaluating reach, effects and cost effectiveness of a mobile health application. The intervention will last for 12 months with follow-up assessments at 3, 6, 9 and 12 months.
Masking Description: Information on the numbers reached will not be masked. All health outcomes are self-reports and self-assessments by the participants and reported in digital surveys. Outcomes will not be influenced by any other outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Safe Step - digital exercise program (Experimental): All included participants will receive full access to the Safe Step application and create their own individual program of strength and balance exercises. During 1 year the participants are recommended to exercise at least 30 minutes, 3 times a week and continuously progress their program. In addition they will every month receive an email with general falls prevention information in a short video.
  Additional support to promote reach and exercise adherence will be provided in the format of technical support and try-out group exercises throughout the recruitment period.
  Interventions: Behavioral: Digital exercise program with support

INTERVENTIONS:
Behavioral: Digital exercise program with support — The Safe Step application includes an instruction movie on how to create and progress an individual exercise program. The exercises, presented in video format, are organized into 10 groups with a main focus on balance (3 groups), lower-limb strength (4 groups), and gait/step (3 groups). The participants choose an exercise suitable for their needs from each group to compose a program of ten exercises.
  Participants use the app to plan their exercises, set reminders, register their exercise, and view statistics. A virtual physiotherapist delivers motivational messages and feed-back. At the end of each month the participants receive an email asking them to report any falls during the past month in a short digital survey. These messages also contains a new video with general falls prevention information.
  Technical support will be provided weekly at senior meeting sites. Try-out group exercises (step 1-3) will be provided by a local wellness association (Friskis&Svettis)

SUMMARY:
The purpose is to evaluate reach, effects and costs effectiveness of a mobile, fall prevention exercise program for older community-dwelling persons (70+ years) in a pragmatic trial.

Information about the study will be spread to the population by letters sent to all households with someone aged 70 years or older, presentations for senior organizations, advertisements on busses, health care centers, senior centers and in social media. Participants will be recruited in one municipality through the website (www.ostersund.se/sakrasteg) including information about the aim and procedures of the study. If seniors themselves judge that they are eligible to participate in the study, they can register by providing their email address. After baseline assessment, through self-reports in a digital survey, participants will get access to the mobile health application. The estimated target group is 2600 persons. Recruitment will be ongoing for six months. The intervention is delivered through the Safe Step application, developed in co-creation with seniors and researchers. Safe Step provides a large repository of evidence-based balance and strength exercises in video formats alongside falls preventive information and advice. With the Safe Step app the user can compose an individualized exercise program suitable for their needs. To help the user adhere to the program a set of behaviour change techniques is provided by the program. The user can set their own goals, get reminders and positive feedback form a virtual physiotherapist, and follow their own progress. Advice on how to integrate the exercises into everyday activities is also offered. The participants will exercise on their own with the help of the application for one year, with a recommendation of 30 minutes at least 3 times/week. In addition, participants will get monthly emails with falls preventive information in short videos, they will also be asked to report any falls by responding to a survey attached to the message.

In order to maximize reach and to support participants to get started using the Safe Step application, technical support and group-based exercise will be provided.

The interventions will last for 1 year with follow up assessments at 3, 6, 9, and 12 months in addition to the monthly fall reports. Effects and cost effectiveness will be evaluated in relation to a previously registered RCT NCT03963570.

ELIGIBILITY:
Inclusion Criteria:

* 70 years or older
* Have fallen or experienced a decline in perceived postural balance during the last year
* Have access to a smartphone or a tablet and uses it regularly
* Have an own email address and uses it
* Ability to understand verbal and written instructions in Swedish
* Can rise from a standard height chair without a person helping
* Independently mobile without a walking aid indoors

Exclusion Criteria:

* Progressive disease where there is likely to be a decline in strength or balance over the next year
* Perceived memory dysfunction that affect everyday life activities
* Taking part in more than 3 hours each week of strenuous physical exercise which makes them out of breath (e.g. dance, gymnastics, gym exercises, running or skiing)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 173 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Reach | 12 months
  The number of participants in relation to estimated size of total target population

SECONDARY OUTCOMES:
Sociodemographic characteristics age | Baseline
  Reach of recruitment will be assessed in relation to age.
Sociodemographic characteristics gender | Baseline
  Reach of recruitment will be assessed in relation to gender.
Sociodemographic characteristics living conditions | Baseline
  Reach of recruitment will be assessed in relation to living conditions).
Functional leg strength | [Time Frame: Change; Baseline, 3 months, 6 months, 9 months, 12 months]
  Self-administered chair stand test (i.e. number of stands during 30 seconds).
Perceived Exertion | Change; Baseline, 3 months, 6 months, 9 months, 12 months
  The Borg Scale of Perceived Exertion during the 30 second chair stand test, rated on a scale between 6 (none) to 20 (maximal exertion).
Self-rated balance | Change; Baseline, 3 months, 6 months, 9 months, 12 months
  Answering the question: "How do you perceive you balance?" on a 5-level ordinal scale ranging from "very good" to "very bad".
Self-rated leg-strength | Change; Baseline, 3 months, 6 months, 9 months, 12 months
  Answering the question: "How do you perceive your leg muscle strength?" on a 5-level ordinal scale ranging from "very good" to "very bad".
Falls efficacy | Change; Baseline, 3 months, 6 months, 9 months, 12 months
  Falls Efficacy Scale-International (FES-I). Concerns about falling is rated for 16 activities (e.g. cleaning the house) on a scale from 1 (not at all concerned ) to 4 (very concerned ). Ratings for each of the 16 activities are summed to a total score ranging from 16 (no concern about falling) to maximum 64 (severe concern about falling)
Health related quality of life | Change; Baseline, 3 months, 6 months, 9 months, 12 months
  Health related quality of life is assessed by the EuroQol 5 dimension 5 level self-report questionnaire (EQ-5D-5L).
  The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression, and a Visual Analogue scale (VAS). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. A 1-digit number express the level selected for each dimension. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state. It should be noted that the numerals 1-5 have no arithmetic properties. The VAS records the respondent's self-rated health on a vertical, visual analogue scale (ranging from 0-100) with endpoints labelled "the best health you can imagine" and "the worst health you can imagine".
Use of the information videos | 3 months, 6 months, 9 months, 12 months
  Answering the question: "Have you watched the videos we sent you by e-mail during the last 3 months?" on a 4-level ordinal scale.
Experienced positive effects of the exercise intervention | 3 months, 6 months, 9 months, 12 months
  Exercise intervention: Self-report of any positive effects of the exercise intervention besides effects on balance and strength. On a nominal scale including an optional text field.
Experienced negative effects of the exercise intervention | 3 months, 6 months, 9 months, 12 months
  Exercise intervention: Self-report of any negative effects (adverse events) of the exercise intervention besides effects on balance and strength. On a nominal scale including an optional text field.
Physical activity | Change: Baseline, 12 months
  Self-reported minutes/week, pre-defined alternatives in 30 minutes blocks up to more than 2 hours.
Exercise adherence throughout the intervention | 12 months
  Adherence to predefined minutes of 3x30 min/week reported continuously through an integrated exercise diary in the Safe step application and by self-report at follow up assessments.
Self-rated improvements in balance | 12 months
  Answering the question: "If you compare with when you started this study a year ago, how would you assess balance today?" on a 5-level ordinal scale on a 5-level ordinal scale ranging from "much better" to "much worse".
Self-rated improvements in leg-strength | 12 months
  Answering the questions: "If you compare with when you started this study a year ago, how would you assess the muscle strength in your legs today?" on a 5-level ordinal scale ranging from "much better" to "much worse".
Rate of attrition | 12 months
  Drop-outs and with-draws in the study
New exercise routines | 12 months
  Participants will be asked if they have started to do any exercises (besides the study intervention) during the intervention period.
Costs related to the interventions | 12 months
  Participants will be asked to report if they have had any cost related to the intervention during the intervention period e.g. for internet access or equipment.
Cost-effectiveness | 12 months
  Cost per falls averted, cost per quality adjusted life years gained.
Participation in technical support sessions | 12 months
  Number of participants participating in technical support sessions
Participation in try-out group exercises | 12 months
  Number of participants participating in try-out group exercise sessions
Fall rate | 12 months
  Falls will be registered every month through a short digital survey, received by email, asking the participant if they had any falls during the last month. If answering yes a few additional questions about when the fall occurred, any resulting injuries and hospital visits will be asked.
Number of fallers | 12 months
  Falls will be registered every month through a short digital survey, received by email, asking the participant if they had any falls during the last month. If answering yes a few additional questions about when the fall occurred, any resulting injuries and hospital visits will be asked.

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Sandlund, Ass Prof, Principal Investigator — Umeå universitet
Locations (1):
- Caring Science Buildning, Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available from the corresponding author on reasonable request.
Access Criteria: Data will be available from the corresponding author on reasonable request. The protocol will be published in an open access journal.

REFERENCES:
- [Derived] Bajraktari S, Zingmark M, Pettersson B, Rosendahl E, Lundin-Olsson L, Sandlund M. Reaching Older People With a Digital Fall Prevention Intervention in a Swedish Municipality Context-an Observational Study. Front Public Health. 2022 Apr 25;10:857652. doi: 10.3389/fpubh.2022.857652. eCollection 2022. PMID 35548075